CLINICAL TRIAL: NCT02456324
Title: A Prospective European Post-Market Clinical Evaluation of the CuraSeal Percutaneous Intraluminal Closure System for Anorectal Fistulas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Curaseal Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP0777
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Anal Fistulas; Rectal Fistulas
Keywords: Fistula, Anorectal
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): Patients Treated with PICS-AF device
  Interventions: Device: PICS-AF Device
- Historical Controls (Other): Patients Treated with Commercially Available Fistula Plug Devices at Same Sites
  Interventions: Device: Historical Controls Treated with Commercially Available Fistula Plugs

INTERVENTIONS:
Device: PICS-AF Device — This is a specialized closure system for anorectal fistulas that is sphincter sparing
  Arms: Treatment Group
Device: Historical Controls Treated with Commercially Available Fistula Plugs — These are patients previously treated with commercially available fistula plugs.
  Arms: Historical Controls

SUMMARY:
The study is designed as a prospective, non-randomized clinical trial comparing safety and effectiveness of the CuraSeal PICS-AF device to historical data from commercially available devices for the treatment of anorectal fistulas.

DETAILED DESCRIPTION:
The primary objective of this post-market study is to generate clinical data to evaluate the performance and safety of the PICS AF devices for the treatment of anorectal fistulas and to compare success rates of fistula closure to historical controls of commercially available devices for anorectal fistula repair performed at the participating clinical sites. Data will be obtained from this study to support the safety and effectiveness of the PICS AF device for promoting fistula closure and healing.

PRIMARY EFFECTIVENESS ENDPOINT:

Fistula closure success at 6 months is defined as complete healing of the fistula tract and associated external opening without drainage or abscess. Fistula closure success for the PICS-AF device will be assessed at the 6 month follow up visit using MRI. The rate of the PICS-AF closure success at 6 months will compared to the closure rate obtained from historical controls that were followed for similar time periods.

PRIMARY SAFETY ENDPOINT:

The proportion of subjects experiencing a serious adverse event (i.e., an infection, enlargement of the fistula, an allergic reaction to the PICS-AF device, etc.) through 6 months of post-procedure follow-up.

SECONDARY ENDPOINTS:

1. Fistula closure at 3 months post-procedure as determined by physical examination.
2. The cessation of egress of enteric fluid from the fistula tract or stable complete closure of the mucosal internal fistula opening by physical examination.
3. Safety post-procedure through 3-month follow-up period.
4. Infection (e.g., systemic or abscess).
5. Time to fistula closure.
6. Need for repeat procedure or other required surgical intervention.
7. Incontinence levels before and after treatment.
8. Quality of life assessments before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent.
2. Subject must be at least 18 years of age and no older than 75 years of age.
3. Subject has been diagnosed with a single internal opening anorectal fistula (not multiple internal openings) that is clinically indicated for treatment.
4. Subject must have a fistula tract that is > 2.0 cm in length based on measurements from imaging studies or upon probing of the fistula tract.
5. Subject should have a clean and infection-free fistula tract that has been properly drained.
6. Subject must be able to comply with study and study follow-up requirements.

Exclusion Criteria:

1. Subject with a life expectancy < 6 months.
2. Subject with anorectal fistula due to Crohn's disease or malignancy.
3. Subject is severely malnourished.
4. Subject with a history of sensitivity or allergy to bovine materials.
5. Subject is on active chemotherapy treatment that may interfere with wound healing.
6. Subject has an active infection (cellulitis) or an undrained abscess in fistula tract.
7. Subject has a horseshoe fistula tract.
8. Subject has a history of radiation therapy to anus or rectum.
9. Subject is affected by uncontrolled diabetes.
10. Subjects with subcutaneous, ano-vaginal, or pouch-vaginal fistula.
11. Subject presents with end stage renal disease requiring dialysis.
12. Subject is pregnant or planning to become pregnant (verbal report).
13. Subject is unable or unwilling to provide informed consent.
14. Subject is currently participating in an investigational drug or another device study that clinically interferes with the current study endpoints.
15. Subject has an American Society of Anesthesia PS classification of greater than 3.
16. Subject is known to be a carrier for drug-resistant bacteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Fistula Closure | 6 months
  Defined as complete healing of the fistula tract and associated external opening without drainage or abscess. Confirmed by MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Hosptial Universitario VIRGEN DEL ROCIO, Seville, Sevilla, Spain